CLINICAL TRIAL: NCT06548672
Title: A Phase Ia/Ib, Open-Label, Dose Escalation and Dose Expansion Study to Evaluate the Safety, Tolerability, Pharmacokinetics (PK), and Preliminary Efficacy of BC3195 in Patients With Locally Advanced or Metastatic Solid Tumors
Brief Title: A Study to Assess the Safety, Pharmacokinetics, and Antitumor Activity of BC3195 in Patients With Advanced or Metastatic Cancer
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Biocity Biopharmaceutics Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: BC3195-102
Record Dates: First submitted 2024-07-11; First posted 2024-08-12 (Actual); Last update posted 2024-08-12 (Actual); Status verified 2024-08

CONDITIONS: Advanced Cancer; Metastatic Solid Tumor
MeSH Terms: conditions — Neoplasm Metastasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Part 1: Phase 1a Dose Escalation (Experimental): Participants will receive BC3195 administered as an intravenous infusion every 3 weeks (Q3W) or according to an alternative dosing regimen, as recommended by the safety monitoring committee (SMC). Multiple dose cohorts will be enrolled. Participants will be monitored for dose limiting toxicities (DLTs) during the DLT assessment period, lasting 21 days. The SMC will determine the recommended phase 2 dose (RP2D) to be administered in Part 2 based on the safety, tolerability, PK, and anti-tumor activity of BC3195
  Interventions: Drug: BC3195
- Part 2: Phase 1b Dose Expansion (Experimental): Participants will receive BC3195 at the RP2D identified in Phase 1a. Approximately 3 to 4 expansion cohorts will be enrolled using a Simon's 2-stage design. Expansion cohorts will focus on tumor types that may derive benefit from BC3195 treatment, including head and neck squamous cell carcinoma (HNSCC), esophageal squamous cell carcinoma (ESCC), breast cancer (BC), non-small cell lung cancer (NSCLC), endometrial cancer (EMC), urothelial cancer (UC), colorectal cancer (CRC), ovarian cancer (OC), pancreatic cancer, and prostate cancer.
  Interventions: Drug: BC3195

INTERVENTIONS:
Drug: BC3195 — BC3195 is a novel antibody drug conjugate (ADC) targeting CDH3 (calcium-dependent adhesion 3). The payload, monomethyl auristatin E (MMAE), is a microtubule disrupting agent covalently attached to the antibody via a cleavable dipeptide linker Val-Cit (vc).

SUMMARY:
This is a phase Ia/Ib, open-label, dose escalation and dose expansion study to evaluate the safety, tolerability, pharmacokinetics, and antitumor activity of BC3195 in subjects with locally advanced or metastatic solid tumors in whom standard treatment has failed (either due to disease progression or intolerance). This study will consist of two parts: Dose escalation (Part 1) and dose expansion (Part 2). Each part will include a screening period, a treatment period, and follow-up period.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients ≥ 18 years of age.
2. Eastern Cooperative Oncology Group (ECOG) performance status of 0-1
3. Subjects with locally advanced or metastatic solid tumors confirmed by histology or cytology who have not benefitted from or are intolerant of available therapy(ies) associated with a reasonable likelihood to confer clinical benefit because of known CDH3 expression, including, albeit not limited to: HNSCC, ESCC, BC, NSCLC, EC, UC, CRC, OC, pancreatic cancer, and prostate cancer.
4. Agree to provide previously archived tumor tissue samples, or newly obtained core biopsy, or excisional biopsy of a previously unirradiated tumor lesion (formalin fixed, paraffin embedded tissue blocks)
5. Subjects with at least one measurable lesion according to RECIST 1.1. Lesions situated in a previously irradiated area are considered measurable if progression has been demonstrated in such lesions
6. Life expectancy ≥ 3 months
7. Subjects with adequate organ function
8. Men or women of childbearing potential must use a highly effective method of contraception during the study and continue to take contraception measures for 6 months after the last dose of the study drug.
9. Patients voluntarily participate in the study and should provide a written informed consent.

Exclusion Criteria:

1. Pregnant or lactating women
2. Prior systemic anticancer treatment, including investigational agents, within 5 half-lives or 4 weeks before the first dose (whichever is shorter)
3. Subjects diagnosed with immunodeficiency within 7 days prior to the first dose of the study drug; or subjects who are receiving longterm systemic steroid therapy or any other form of immunosuppressive therapy
4. Previously received allogeneic tissue/solid organ transplantation
5. Patients who have received radiation therapy within 2 weeks prior to the start of study treatment or with a history of radiation pneumonitis.
6. Known active CNS metastases and/or cancerous meningitis. Subjects with previously treated brain metastases who meet the following conditions are permitted to participate in the study: radiologically stable, that is, repeat imaging shows no evidence of progression for at least 4 weeks, clinically stable, and no steroid therapy is required for at least 14 days prior to the first dose of study treatment
7. Active viral infection requiring systemic therapy during the screening period
8. Clinically uncontrolled pericardial effusion, pleural effusion, or ascites at screening
9. Has a history of (non-infectious) pneumonitis / interstitial lung disease that required steroids or has current pneumonitis / interstitial lung disease
10. Hypertension that cannot be well-controlled with medical treatment. Not well-controlled is defined as systolic blood pressure >150 mmHg or diastolic blood pressure >90 mmHg (adjustment of hypertensive medication prior to study initiation is permitted, but the mean of the most recent three consecutive blood pressure records prior to study entry must be ≤150/90 mmHg [with at least 2- minute interval between each measurement])
11. Cardiovascular disease of clinical significance: Including New York Heart Association [NYHA] Class II-IV, congestive heart failure, second-degree or higher heart block, myocardial infarction within the past 3 months, unstable arrhythmia or unstable angina, marked QT interval prolongation (12-lead ECG showing baseline-corrected QTc interval >480 ms), cerebral infarction within 3 months, or having received PTCA or CABG within 6 months
12. Subjects with active or chronic corneal disorders, with other active ocular conditions requiring ongoing therapy or with any clinically significant corneal disease that prevents adequate monitoring of drug-induced keratopathy
13. Grade 2 or higher peripheral neuropathy. Other toxicities caused by prior anti-tumor therapy has not recovered to ≤ grade 1 (per CTCAE 5.0) (except for alopecia, pigmentation, and other events judged by the Investigator to be tolerable) or the level specified by the inclusion/exclusion criteria in this study
14. Subjects with any active infection that requires anti-infective therapy judged by the investigators
15. Known hypersensitivity or delayed hypersensitivity reactions to the same class and/or any components of BC3195
16. Subjects who received strong CYP3A4 inhibitors and Strong CYP3A4 inducers within 14 days or 5 half-lives whichever is shorter, before the first dose (refer to Appendix 7 for a list of strong CYP3A4 inhibitors and inducers)
17. Subjects are not suitable for participating the study judged by the investigators
18. Subjects with poor compliance, who are unwilling to or unable to follow study procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 148 (Estimated)
Dates: Start 2024-06-24 (Actual); Primary Completion 2027-04-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of Dose Limiting Toxicities (DLTs) | First 21 days of treatment
Determination of the Maximum Tolerated Dose (MTD) and/or Recommended Phase 2 Dose (RP2D) | Day 1 of treatment through 30 days after the last dose
Incidence and Severity of All Adverse Events (AEs) | Screening through 12 weeks after the last dose

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | Day 1 of treatment through 6 weeks after the last dose
  Assessed according to the Response Evaluation Criteria in Solid Tumors (RECIST) V1.1
Disease Control Rate (DCR) | Day 1 of treatment through 6 weeks after the last dose
  Proportion of subjects with CR, PR, and stable disease (SD)
Duration of Response (DoR) | Day 1 of treatment through 6 weeks after the last dose
  Defined as the time from the date when the measurement criteria were met for complete or partial response (whichever occurred first) until the date of the first observed PD or death of any cause
Time to Progression (TTP) | Day 1 of treatment through 6 weeks after the last dose
  Defined as the length of time from the start of treatment until first evidence of disease progression
Progression Free Survival (PFS) | Day 1 of treatment through 6 weeks after the last dose
  Defined as the time from which the subject is enrolled to the date of any recorded disease progression or the death of any cause
Overall Survival (OS) | Patient consent until death Day 1 of dosing until the date of death from any cause assessed up to 100 months
  Defined as the time from Day 1 of dosing until the date of death from any cause assessed up to 100 months
Area under the curve (AUC) of BC3195 | Day 1 of dosing through 21 days post last dose
  Area under the BC3195 time vs concentration curve
Maximum concentration (Cmax) of BC3195 | Day 1 of dosing through 21 days post last dose
  Maximum concentration observed following dosing
Time to reach maximum concentration (Tmax) of BC3195 | Day 1 of dosing through 21 days post last dose
  Time at which the maximum concentration of BC3195 is observed
Half-life (t 1/2) of BC3195 | Day 1 of dosing through 21 days post last dose
  Time at which BC3195 concentration is reduced by one half
Volume of distribution (Vd) of BC3195 | Day 1 of dosing through 21 days post last dose
  Volume of distribution
Clearance (CL) of BC3195 | Day 1 of dosing through 21 days post last dose
  Volume of drug cleared in a period of time
Immunogenicity indicators | Day 1 of dosing through 30 days post last dose
  Anti-drug antibody (ADA)

CONTACTS AND LOCATIONS:
Locations (1):
- Case Western Reserve University, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No